CLINICAL TRIAL: NCT00554866
Title: Carbamoyl-phosphate Synthase Gene Polymorphisms Influencing Plasma L-arginine Concentrations in Preterm Infants
Brief Title: L-arginine Concentrations and CPS Polymorphisms in VLBW Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 07-2-018
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Infant, Very Low Birth Weight
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VLBW between 6 and12 hours after birth (Experimental): Blood sample and buccal swab sample. One blood sample (500 mL) will be obtained from each VLBW infant between 6 and12 hours after birth from an umbilical-artery or peripheral artery catheter.
  Additional DNA collection buccal cell samples were obtained with a sterile OmniSwab.
  Interventions: Other: blood sample and buccal swab sample

INTERVENTIONS:
Other: blood sample and buccal swab sample — one blood sample (500 mL) will be obtained from each VLBW infant between 6 and12 hours after birth from an umbilical-artery or peripheral artery catheter.
  Additional DNA collection buccal cell samples were obtained with a sterile OmniSwab.
  Other Names: OmniSwab

SUMMARY:
Plasma L-arginine concentrations are decreased in premature infants with necrotizing enterocolitis (NEC). A carbamoyl-phosphate synthetase 1 (CPS1) polymorphism has been correlated with low plasma concentrations of L-arginine in neonates (> 35 weeks of gestation). Recently Moonen et al (Pediatr Res 2007; 62(2):188-90) described a correlation between this CPS1 T1405N single nucleotide polymorphism (SNP) and the presence of NEC in VLBW infants. However there is no data about the correlation between the plasma arginine concentrations and the T1405N SNP in the CPS-1 gene in VLBW infants. In the present project we postulate that T1405N SNP in the CPS-1 gene is associated with lower plasma arginine concentrations and is also a risk factor for the development of NEC.

DETAILED DESCRIPTION:
Plasma L-arginine concentrations are decreased in premature infants with necrotizing enterocolitis (NEC). A C-to-A nucleotide transversion (T1405N) in the gene that encodes carbamoyl-phosphate synthetase 1 (CPS1), the rate-limiting enzyme in the urea cycle, has been correlated with low plasma concentrations of L-arginine in neonates (> 35 weeks of gestation). Recently Moonen et al (Pediatr Res 2007; 62(2):188-90) described a correlation between this CPS1 T1405N single nucleotide polymorphism (SNP) and the presence of NEC in VLBW infants. However there is no data about the correlation between the plasma arginine concentrations and the T1405N SNP in the CPS-1 gene in VLBW infants. In the present project we postulate that T1405N SNP in the CPS-1 gene is associated with lower plasma arginine concentrations and is also a risk factor for the development of NEC.

ELIGIBILITY:
Inclusion Criteria:

* VLBW infants (< 30 weeks and < 1500 gram birth weight).

Exclusion Criteria:

* Blood transfusion, enteral or parenteral protein intake, or inhaled nitric oxide administration before time of the blood sample (obtained between 6 and 12 hours after birth).
* Parents not able to give informed consent.

Ages: 6 Hours to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 477 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the association between the T1405N SNP in the CPS-1 gene and lower plasma L-arginine concentrations | 2 years

SECONDARY OUTCOMES:
To determine whether the T1405N SNP in the CPS-1 gene is associated with a higher risk of NEC | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Villamor, MD, PhD, Principal Investigator — Maastricht University Hospital
Locations (4):
- Italy (2):
  - Carlo Poma Hospital, Mantova
  - Cattedra di Neonatologia-Università degli Studi di Milano, Milan
- Maastricht University Hospital, Maastricht, Limburg, Netherlands
- Complejo Universitario Hospitalario Insular-Materno Infantil, Las Palmas de Gran Canaria, Spain